CLINICAL TRIAL: NCT06171802
Title: EMPagliflozin After Aortic Valve Replacement - The EMPAVR Study - A Randomized Clinical Trial
Brief Title: EMPagliflozin After Aortic Valve Replacement
Acronym: EMPAVR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Emil Loldrup Fosbol, Professor, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-504731-40-01
Record Dates: First submitted 2023-11-23; First posted 2023-12-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-11

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; Aortic Valve Replacement; Transcatheter Aortic Valve Implantation; Aortic Valve; Sodium-Glucose Cotransporter-2 inhibitor; SGLT2i; Empagliflozin
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Active Comparator): Empagliflozin 1 capsule of 10 mg, once daily for six months.
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): 1 capsule of placebo, once daily for six months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — 10 mg empagliflozin daily for six months
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — Placebo capsule once daily for six months
  Arms: Placebo

SUMMARY:
The study is a randomized, placebo-controlled, and double-blinded trial in patients with aortic stenosis (AS) undergoing aortic valve replacement (AVR). After AVR, patients will be randomized 1:1 to empagliflozin (SGLT2i) or placebo to investigate whether empagliflozin is superior to placebo in reducing left ventricular mass and improve symptoms to 6 months.

DETAILED DESCRIPTION:
In this randomized, placebo-controlled, and double-blinded trial we investigate whether empagliflozin (SGLT2i) is superior to placebo in reducing left ventricular mass and improve symptoms.

All patients with AS who are referred to Rigshospitalet for AVR (both surgical and transcatheter approaches) will be screened for in- and exclusion criteria in the medical record based on the Danish Health Act §46 by the PI, co-PI, or a delegated study nurse. If the patient fulfills the inclusion criteria and none of the exclusions criteria, the patient is invited to participate in the study.

Included patients will be randomized 1:1 in blocks of 2, 4, and 6 patients to either Empagliflozin 10 mg daily or placebo. Point of randomization will be in the hospital when the patients has undergone AVR.

The total treatment period is 6 months with either 10 mg Empagliflozin or placebo. The trial participants will receive conventional treatment, which will be carried out irrespective of the inclusion in the trial in accordance with national guidelines. Routine clinical check-ups irrespective of the trial setup will be performed at 3 months after discharge, and study-outcomes will be assessed at discharge, 3 months, and 6 months (eg. echocardiography). Blood samples (including N-Terminal-proBNP, renal function and electrolytes, hemoglobin and HbA1c) will be part of such routine visits as well as a standardized symptom-scoring tool (KCCQ and NYHA classification). Compliance will be evaluated at 1-, 3- and 6-months. The assessment for 1-month will be per telephone and the assessment at 3- and 6-months will be at the routine clinical check-ups in the outpatient clinic.

The CT scan performed in the planning of the procedure will be used for the baseline assessment (before AVR). An identical exam (CT scan) will be performed at 6 months to assess change in LV mass.

ELIGIBILITY:
Inclusion Criteria:

Severe symptomatic aortic stenosis AND Surgical or transcatheter aortic valve replacement within 14 days

Exclusion Criteria:

* Prior treatment with a SGLT2i
* Left ventricular ejection fraction < 45%
* Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min
* Hypersensitivity to empagliflozin or placebo tablet
* Type I Diabetes
* Patients who do not understand Danish or English
* Women who are pregnant or are nursing or plan to become pregnant during trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular mass indexed to body surface area | 6 months from discharge post-Aortic Valve Replacement
  Change in left ventricular mass indexed to body surface area (measured by CT) from pre-Aortic Valve Replacement to 6-months post-Aortic Valve Replacement

SECONDARY OUTCOMES:
LVESVi | 6-months from discharge post-aortic valve replacement
  Left ventricular end-systolic volume indexed to body surface (LVESVi) (measured by CT)
LV GLS (echo) | 3- and 6-months from discharge
  Left ventricular global longitudinal strain (LV GLS) (measured by echocardiography)
N-terminal pro B-type natriuretic peptide (NT-proBNP) change | 3- and 6-months from discharge
  NT-proBNP change from baseline to 6 months
Death and readmission for any non-planned cause | 6 months from discharge date (after aortic valve replacement)
  A composite outcome of death and readmission for any non-planned cause
Death | 6 months from discharge date (after aortic valve replacement)
  Death during follow-up, from discharge to 6-months after discharge
Readmission for any cause | 6 months from discharge date (after aortic valve replacement)
  Readmission for any cause to any hospital after discharge
Admission for heart failure | 6 months from discharge date (after aortic valve replacement)
  Admission for heart failure to any hospital
Kansas City Cardiomyopathy Questionaire (KCCQ) | 6 months from discharge date (after aortic valve replacement)
  Change in symptom score (KCCQ) at 6-months. KCCQ scores are scaled from 0 to 100, where scores represent health status as follows: 0-24: very poor to poor; 25-49: poor to fair; 50-74: fair to good; and 75-100: good to excellent.
  In this study a change of 5 points is considered a meaningful change.
Quality of Life (QoL) - The Minnesota Living with Heart Failure Questionnaire (MLHFQ) | 6 months from discharge date (after aortic valve replacement)
  Quality of life assessment at baseline and 6 months after discharge post-AVR using the Minnesota Living with Heart Failure Questionnaire (MLHFQ).
  MLHFQ consist of 21 questions. The response format ranges from 0 (none or not applicable), to 1 (very little) to 5 (very much). The sum of responses ranges from 0 to 105. The score increases with adverse impact of the disease on the respondent's life.
New York Heart Association (NYHA) Functional Classification | 3- and 6-months from discharge date (after aortic valve replacement)
  Change in symptom score at 6 months (NYHA classification).
  The NYHA classification places patients in one of four categories based on limitations of physical activity. Class I: No limitation of physical activity; Class II: Slight limitation of physical activity; Class III: Marked limitation of physical activity; Class IV: Symptoms of heart failure at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Emil L. Fosbøl, MD, PhD, Principal Investigator — University Hospital of Copenhagen - Rigshospitalet
Locations (1):
- University Hospital of Copenhagen, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No